CLINICAL TRIAL: NCT01918020
Title: Impact Study of Minnesota SNAP-Ed Health and Nutrition Education Programs
Acronym: SNAP-Ed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1206S15445
Record Dates: First submitted 2013-07-26; First posted 2013-08-07 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Obesity; Child
Keywords: Fruit; Vegetables; Motor Activity
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Fruit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Go Wild with Fruits and Veggies! (Experimental): This group will receive nutrition education to learn about fruits and vegetables and physical activities right from the start of the experiment.
  Interventions: Behavioral: Go Wild with Fruits and Veggies!
- Go Wild with Fruits and Veggies! delayed (Other): This group will only receive nutrition education about 4 months after the experiment starts.
  Interventions: Behavioral: Go Wild with Fruits and Veggies! delayed

INTERVENTIONS:
Behavioral: Go Wild with Fruits and Veggies! — Fruits and Vegetables
  Arms: Go Wild with Fruits and Veggies!
Behavioral: Go Wild with Fruits and Veggies! delayed — Go Wild with Fruits and Veggies! delayed
  Arms: Go Wild with Fruits and Veggies! delayed

SUMMARY:
Supplemental Nutrition Assistance Program - Education (SNAP-Ed) is a national initiative with the goal of improving the health and wellbeing of low income families. University of Minnesota Extension every year offers nearly 4000 educational events, serving approximately 70,000 Minnesotans through the program. Extension is conducting an impact study to determine program effectiveness and assess sustained changes of participants and their families that can be directly attributed to programming on a larger and methodically sound scale.

ELIGIBILITY:
Inclusion Criteria:

* Third grade elementary students
* Schools that are eligible for SNAP ED funding (have more than 50% students received free/reduced lunch)

Exclusion Criteria:

* Other grade elementary students
* Schools that are not eligible for SNAP ED funding

Ages: 8 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 796 (Actual)
Dates: Start 2012-09; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To assess changes in adiposity level among the program participants indicated by BMI measurements. | We will assess BMI in the 1st, 3rd, 5th and 12th month
  We assess BMI of participants by using standardized stadiometers and weighing scales to attain weights and heights. Birthdates and sex of program participants were also acquired. Then, using the information of their birthdates, weight and heights, BMI percentile and BMI will be computed and analyzed.

SECONDARY OUTCOMES:
To assess changes of fruit and vegetable intake and among program participants. | We will measure the changes of fruits and vegetable intakes in the 1st month (baseline), 3rd month, 7th month, and 12th month
  We use fruits and vegetables frequency retrospective questions and "A day in the life" survey to assess the fruits and vegetable intake. Composite values of these two measures will decide the levels of changes in intakes.
To assess changes of physical activity levels among program participants. | We will measure the changes of physical activity level in the 1st month (baseline), 3rd month, 7th month, and 12th month
  We use Yamax Digiwalker (SW700) pedometer, physical activity questions, and parent proxy surveys to assess the physical activity levels. Composite values of all measures will be computed to determine the levels of change.

CONTACTS AND LOCATIONS:
Overall Officials: G. Ali Hurtado, Doctorate, Principal Investigator — University of Minnesota Extension Center for Family Development
Locations (1):
- University of Minnesota Extension Center for Family Development, Saint Paul, Minnesota, United States